CLINICAL TRIAL: NCT06030414
Title: A Phase 1, Single-site, Open-label Study to Determine the Safety and Tolerability of Single and Multiple Doses of Intranasally Administered LMN-301 in Healthy Volunteers
Brief Title: A Study to Determine the Tolerability of Intranasal LMN-301
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: COV01
Record Dates: First submitted 2023-08-10; First posted 2023-09-11 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sentinel Cohort (Experimental)
  Interventions: Biological: LMN-301
- Main Cohort Group 1 (Experimental)
  Interventions: Biological: LMN-301
- Main Cohort Group 2 (Experimental)
  Interventions: Biological: LMN-301
- Main Cohort Group 3 (Experimental)
  Interventions: Biological: LMN-301

INTERVENTIONS:
Biological: LMN-301 — Intranasally administered powder.

SUMMARY:
LMN-301 is to prevent infection by severe acute respiratory syndrome-corona virus (SARS-CoV-2) (the virus causing coronavirus disease of 2019 (COVID-19) in uninfected individuals. This study aims to assess whether the formulation will cause irritation when administered in the nose, and how long its protective effects will last.

Thirty five healthy adult volunteers will participate in this study.

ELIGIBILITY:
Individuals must meet all the following criteria to be eligible to participate in this study:

1. Adult (between 18 and 65 years of age) at screening
2. BMI ≥ 18.0 and ≤ 30.0 kg/m2, with a maximum body weight of 120 kg at screening.
3. General good health, without significant medical illness or abnormal physical examination findings per investigator discretion.
4. No clinically significant laboratory values at screening for haematology, serum chemistry, coagulation, and urinalysis in the opinion of the Investigator. A repeat test is allowed at the investigator's discretion.
5. Normal electrocardiogram (ECG) with no QTcF prolongation.
6. Must have provided written informed consent to participate in the clinical trial before any study-related activities are carried out and, in the Investigator's opinion, must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
7. In the investigator's opinion, participant is willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Female volunteers:

1. Must be of non-child-bearing potential, i.e., surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause (confirmed with follicle stimulating hormone (FSH) testing), or
2. If of child-bearing potential, must have a negative serum pregnancy test at screening and negative urine pregnancy test before the first study drug administration. They must agree not to attempt to become pregnant, must not donate ova, and must agree to use a highly effective method of contraception from signing consent, throughout the study and for at least 30 days after the last dose of study drug. For contraception guidelines see Appendix 4.

   9. Male volunteers must agree not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use a condom in addition to having the female partner use a highly effective contraceptive method (Appendix 4) from signing consent, during the study, and at least 90 days after the last dose of study drug.

   Exclusion Criteria

   Individuals will be excluded from this study if they meet any of the following criteria:
   1. History or presence of clinically significant disease, including (but not limited to) clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological or psychiatric disease, including any acute illness or surgery within the past 3 months prior to screening determined by the PI to be clinically relevant.
   2. Known allergy or previous anaphylaxis to any components of the investigational product
   3. Allergies, history of allergic disease or chronic respiratory diseases including mild asthma. History of childhood asthma or childhood allergies are not exclusionary.
   4. History of nasal or upper respiratory pathology or abnormalities
   5. Ongoing, defined as within 30 days of dosing through end of follow-up, usage of nasal spray or nasal drops
   6. Treatment with an experimental device or compound within 30 days of the first dose of study drug.
   7. Treatment within 30 days of the first dose of the study medication or planned use within the study period with immunomodulator or immunosuppressant agent or medicines over-the-counter (OTC), herbal, prescription, or supplement) with significant activity in the respiratory tract.
   8. Pregnancy, anticipated pregnancy, or breastfeeding/lactating
   9. Alcohol or drug abuse/dependency (defined as more than 10 standard drinks per week or more than 4 standard drinks on any one day, where 1 standard drink is 10 g of pure alcohol) within 3 months prior to screening.
   10. Positive urine toxicology screen for drugs of abuse. Repeat testing is allowed at investigator discretion. Tobacco or nicotine consumption is not permitted from screening and until the end of follow-up.
   11. Positive alcohol breath test. Repeat test is allowed at investigator discretion.
   12. Individuals unable or unwilling to provide adequate informed consent
   13. COVID-19 positive
   14. Positive test results for active human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Cohort: Part A: single fixed dose of 50 mg LMN-301 IN (25 mg in each nostril)
- Main Cohort Group 1: Cohort 2, Part B: 50 mg (25 mg in each nostril) LMN-301 once every third day for 12 days (4 doses total)
- Main Cohort Group 2: Cohort 2, Part B: 50 mg (25 mg in each nostril) once every other day for 12 days (6 doses total)
- Main Cohort Group 3: Cohort 2, Part B: Part B: 50 mg (25 mg in each nostril) once every day for 12 days (12 doses total)
Period: Overall Study
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Started | 5 | 10 | 10 | 10
Completed | 5 | 10 | 9 | 10
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Healthy adult volunteers aged 19-65, with BMI between 18.0 and 30.0 kg/m, and a maximum body weight of 120 kg.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3 | Total
Number analyzed (Participants) | 5 | 10 | 10 | 10 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 10 | 10 | 35
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (15.66) | 40.6 (16.32) | 37.9 (14.63) | 33.8 (14.33) | 37.4 (14.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 6 | 2 | 15
  Male | 2 | 6 | 4 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 3 | 5
  Not Hispanic or Latino | 5 | 9 | 9 | 7 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 1 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 3 | 6 | 8 | 5 | 22
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 10 | 10 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: All adverse events (AEs) will be coded using the latest version of MedDRA by system organ class (SOC) and preferred term, classified from verbatim terms. The number of treatment-emergent AEs (TEAEs) as well as the number and percentage of participants with at least one TEAE, will be summarized by SOC and preferred term. Summaries of TEAEs by severity as assessed by CTCAE v5.0 and relationship will also be presented. Summaries will also be presented for serious adverse events (SAEs), TEAEs leading to death or study withdrawal. The duration of all AEs will be determined and included in the listings. Solicited and unsolicited TEAEs will be summarized separately.
Time Frame: Daily for 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 10 | 10
Participants | 5 | 9 | 10 | 8

2. Primary Outcome: Number of Participants Discontinuing From the Study
Description: The endpoint is the number of participants discontinuing from the study.
Time Frame: For 28 days after the first dose of LMN-301
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 10 | 10
Participants | 0 | 0 | 1 | 0

3. Primary Outcome: Changes From Baseline of Systolic and Diastolic Blood Pressure.
Description: Changes from baseline for systolic and diastolic blood pressure will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: In part A vital signs are measured on Days 1 (4 timepoints), 2, 8 and 14. In part B vital signs are measured on Days 1 (3 timepoints), 3 or 4, 7, 10 or 11, 14 and 28.
Population: Healthy volunteers aged 18-65 years, BMI between 18.0 and 30.0 kg/m, and a maximum body weight of 120 kg.
Measure: Mean (Standard Deviation); unit: Delta from baseline blood pressure(mmHg)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Delta from baseline blood pressure(mmHg)
  Change from baseline in systolic blood pressure (mmHg) - Day 1, 0.25 hour post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 1, 0.25 hour post-dose |  | 1.4 (11.21) | -1.3 (8.22) | -2.4 (4.50)
  Change from baseline in systolic blood pressure (mmHg) - Day 1, 0.5 hour post-dose | 0.4 (8.08) | -1.7 (10.13) | -2.8 (7.02) | -2.5 (10.81)
  Change from baseline in systolic blood pressure (mmHg) - Day 1, 1 hour post-dose | -1.8 (8.58) | -1.9 (9.88) | -2.2 (5.39) | -0.9 (5.11)
  Change from baseline in systolic blood pressure (mmHg) - Day 1, 4 hours post-dose | 5.2 (6.61) | 4.7 (8.53) | -1.1 (6.33) | 1.2 (7.07)
  Change from baseline in systolic blood pressure (mmHg) - Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in systolic blood pressure (mmHg) - Day 2 | -0.6 (8.32) |  |  |
  Change from baseline in systolic blood pressure (mmHg) - Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 3 |  | 0 (0) | -4.3 (6.33) | -1.5 (9.00)
  Change from baseline in systolic blood pressure (mmHg) - Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 4 |  | -1.6 (10.56) | 0 (0) | 0 (0)
  Change from baseline in systolic from baseline in blood pressure (mmHg) - Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic from baseline in blood pressure (mmHg) - Day 7 |  | 2.9 (14.13) | -3.8 (8.51) | -4.1 (7.00)
  Change from baseline in systolic change from baseline in blood pressure (mmHg) - Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in systolic change from baseline in blood pressure (mmHg) - Day 8 | 0.4 (15.92) |  |  |
  Change from baseline in systolic blood pressure (mmHg) - Day 10: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 10 |  | 1.3 (11.68) | 0 (0) | 0 (0)
  Change from baseline in systolic blood pressure (mmHg) - Day 11: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 11 |  | 0 (0) | -6.6 (8.65) | -2.9 (6.92)
  Change from baseline in systolic blood pressure (mmHg) - Day 14 | 1.2 (7.79) | 3.4 (15.06) | -4.0 (9.23) | -1.5 (8.96)
  Change from baseline in systolic blood pressure (mmHg) - Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in systolic blood pressure (mmHg) - Day 28 |  | 1.6 (14.80) | -3.1 (7.56) | 2.2 (8.57)
  Change from baseline in diastolic blood pressure (mmHg) - Day 1, 0.25 hour post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 1, 0.25 hour post-dose |  | 0.2 (6.11) | -0.6 (3.91) | 0.3 (6.60)
  Change from baseline in diastolic blood pressure (mmHg) - Day 1, 0.5 hour post-dose | 2.2 (4.76) | -2.7 (5.87) | -2.0 (4.78) | -1.8 (6.37)
  Change from baseline in diastolic blood pressure (mmHg) - Day 1, 1 hour post-dose | 1.0 (7.21) | -1.9 (5.09) | -1.8 (5.18) | 0.9 (6.26)
  Change from baseline in diastolic blood pressure - Day 1, 4 hours post-dose | 1.0 (10.32) | -2.1 (5.99) | -2.5 (5.66) | -0.4 (7.88)
  Change from baseline in diastolic blood pressure (mmHg) - Day 2 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in diastolic blood pressure (mmHg) - Day 2 post-dose | 0.0 (4.18) |  |  |
  Change from baseline in diastolic blood pressure (mmHg) - Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 3 |  | 0 (0) | -3.4 (7.47) | -1.9 (6.56)
  Change from baseline in diastolic blood pressure (mmHg) - Day 4 | 0 (0) | 0.1 (7.31) | 0 (0) | 0 (0)
  Change from baseline in diastolic blood pressure (mmHg) - Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 7 |  | -0.3 (7.09) | -3.9 (8.88) | -1.1 (4.72)
  Change from baseline in diastolic blood pressure (mmHg) - Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in diastolic blood pressure (mmHg) - Day 8 | -1.6 (4.39) |  |  |
  Change from baseline in diastolic blood pressure (mmHg) - Day 10: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 10 |  | 0.9 (8.51) | 0 (0) | 0 (0)
  Change from baseline in diastolic blood pressure (mmHg) - Day 11: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 11 |  | 0 (0) | -6.0 (7.40) | -0.7 (6.99)
  Change from baseline in diastolic blood pressure (mmHg) - Day 14 | 1.6 (5.77) | 1.4 (9.79) | -2.2 (5.70) | 0.7 (6.63)
  Change from baseline in diastolic blood pressure (mmHg) - Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in diastolic blood pressure (mmHg) - Day 28 |  | 0.0 (8.33) | -3.1 (7.25) | 4.1 (6.19)

4. Primary Outcome: Changes From Baseline of Pulse Rate.
Description: Changes from baseline for pulse rate will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: as for outcome 3
Population: Healthy volunteers aged 18-65 years, BMI between 18.0 and 30.0 kg/m, and a maximum body weight of 120 kg.
Measure: Mean (Standard Deviation); unit: Change from baseline of pulse rate
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Change from baseline of pulse rate
  Change from baseline in pulse rate (beats/min ) - Day 1, 0.25 hour post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 1, 0.25 hour post-dose |  | -4.2 (7.51) | -5.0 (3.32) | -3.0 (4.11)
  Change from baseline in pulse rate (beats/min ) - Day 1, 0.5 hour post-dose | -4.8 (3.27) | -5.4 (6.40) | -4.6 (2.99) | -4.0 (5.98)
  Change from baseline in pulse rate (beats/min ) - Day 1, 1 hour post-dose | -7.0 (1.87) | -3.0 (8.70) | -4.0 (4.59) | -5.0 (5.08)
  Change from baseline in pulse rate (beats/min ) - Day 1, 4 hours post-dose | 1.4 (2.70) | 3.1 (7.80) | 3.1 (4.23) | 2.6 (7.21)
  Change from baseline in pulse rate (beats/min ) - Day 2 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in pulse rate (beats/min ) - Day 2 post-dose | 3.4 (7.27) |  |  |
  Change from baseline in pulse rate (beats/min ) - Day 3 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 3 post-dose |  | 0 (0) | 2.7 (7.12) | -1.8 (4.21)
  Change from baseline in pulse rate (beats/min ) - Day 4 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 4 post-dose |  | -0.5 (6.26) | 0 (0) | 0 (0)
  Change from baseline in pulse rate (beats/min ) - Day 7 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 7 post-dose |  | 5.0 (10.12) | 8.3 (8.29) | 0.8 (8.05)
  Change from baseline in pulse rate (beats/min ) - Day 8 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in pulse rate (beats/min ) - Day 8 post-dose | 3.4 (8.29) |  |  |
  Change from baseline in pulse rate (beats/min ) - Day 10 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 10 post-dose |  | 5.4 (11.1) | 0 (0) | 0 (0)
  Change from baseline in pulse rate (beats/min ) - Day 11 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 11 post-dose |  | 0 (0) | 6.3 (4.85) | -2.0 (3.33)
  Change from baseline in pulse rate (beats/min ) - Day 14 post-dose | 4.6 (8.32) | 3.2 (7.22) | 6.7 (6.02) | 2.3 (2.36)
  Change from baseline in pulse rate (beats/min ) - Day 28 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in pulse rate (beats/min ) - Day 28 post-dose |  | 1.5 (6.67) | -1.4 (5.96) | -1.5 (7.31)

5. Primary Outcome: Changes From Baseline of Oral Temperature.
Description: Changes from baseline for oral temperature will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: as for outcome 3
Population: Healthy volunteers aged 18-65 years, BMI between 18.0 and 30.0 kg/m, and a maximum body weight of 120 kg.
Measure: Mean (Standard Deviation); unit: Change from baseline of temperature (°C)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Change from baseline of temperature (°C)
  Change from baseline in temperature (°C) - Day 1, 0.25 hour post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 1, 0.25 hour post-dose |  | -0.15 (0.381) | -0.04 (0.388) | 0.13 (0.347)
  Change from baseline in temperature Change from baseline in (°C) - Day 1, 0.5 hour post-dose | -0.42 (0.476) | 0.01 (0.185) | -0.1 (0.613) | 0.17 (0.460)
  Change from baseline in temperature (°C) - Day 1, 1 hour post-dose | -0.42 (0.228) | -0.11 (0.805) | -0.02 (0.322) | 0.14 (0.327)
  Change from baseline in temperature (°C) - Day 1, 4 hour post-dose | -0.10 (0.418) | 0.13 (0.313) | -0.34 (0.488) | 0.16 (0.422)
  Change from baseline in temperature (°C) - Day 2 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in temperature (°C) - Day 2 post-dose | -0.34 (0.297) |  |  |
  Change from baseline in temperature (°C) - Day 3 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 3 post-dose |  | 0 (0) | -0.25 (0.788) | 0.18 (0.368)
  Change from baseline in temperature (°C) - Day 4 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 4 post-dose |  | -0.8 (0.437) | 0 (0) | 0 (0)
  Change from baseline in temperature (°C) - Day 7 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 7 post-dose |  | -0.18 (0.338) | -0.10 (0.424) | 0.27 (0.350)
  Change from baseline in temperature (°C) - Day 8 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in temperature (°C) - Day 8 post-dose | -0.34 (0.658) |  |  |
  Change from baseline in temperature (°C) - Day 10 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 10 post-dose |  | -0.17 (0.374) | 0 (0) | 0 (0)
  Change from baseline in temperature (°C) - Day 11 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 11 post-dose |  | 0 (0) | -0.10 (0.274) | 0.17 (0.353)
  Change from baseline in temperature (°C) - Day 14 post-dose | -0.32 (0.653) | -0.22 (0.424) | 0.02 (0.549) | 0.33 (0.472)
  Change from baseline in temperature (°C) - Day 28 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in temperature (°C) - Day 28 post-dose |  | -0.18 (0.394) | -0.39 (0.446) | 0.25 (0.517)

6. Primary Outcome: Changes From Baseline of Hemoglobin.
Description: Clinical laboratory safety data will be summarized by laboratory measures like hemoglobin. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: There are timepoints for sentinel cohort Part A that were not collected for main cohort Part B; because of this there are some timepoint collections listed as "0" subjects analyzed for that particular timepoint. Otherwise "0" has been entered where data was not collected for that timepoint.
Measure: Mean (Standard Deviation); unit: Changes from baseline of hemoglobin(g/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Changes from baseline of hemoglobin(g/L)
  Change from baseline in hemoglobin (g/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in hemoglobin (g/L) Day 2 | 2.6 (10.04) |  |  |
  Change from baseline in hemoglobin (g/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hemoglobin (g/L) Day 3 |  | 0 (0) | -2.8 (7.07) | -1.3 (6.50)
  Change from baseline in hemoglobin (g/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hemoglobin (g/L) Day 4 |  | -1.5 (7.12) | 0 (0) | 0 (0)
  Change from baseline in hemoglobin (g/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hemoglobin (g/L) Day 7 |  | -0.6 (4.28) | -9.3 (5.36) | -4.7 (6.25)
  Change from baseline in hemoglobin (g/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in hemoglobin (g/L) Day 8 | -0.8 (7.79) |  |  |
  Change from baseline in hemoglobin (g/L) Day 14 | -2.2 (11.08) | -3.2 (5.45) | -5.4 (5.17) | -3.8 (7.22)
  Change from baseline in hemoglobin (g/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hemoglobin (g/L) Day 28 |  | -4.7 (5.77) | -4.9 (9.44) | -2.7 (6.53)

7. Primary Outcome: Changes From Baseline of Respiratory Rate.
Description: Changes from baseline for respiratory rate will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: In part A respiratory rate is measured on Days 1 (4 timepoints), 2, 8 and 14. In part B vital signs are measured on Days 1 (3 timepoints), 3 or 4, 7, 10 or 11, 14 and 28.
Population: Healthy volunteers aged 18-65 years, BMI between 18.0 and 30.0 kg/m, and a maximum body weight of 120 kg.
Measure: Mean (Standard Deviation); unit: Respiratory rate (breaths per minute)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Respiratory rate (breaths per minute)
  Change from baseline in respiratory rate (breaths/minute) - Day 1, 0.25 hours post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 1, 0.25 hours post-dose |  | -0.5 (2.88) | -3.1 (2.67) | -0.3 (1.16)
  Change from baseline in Respiratory Rate (breaths/minute) - Day 1, 0.5 hour post-dose | -3.6 (2.19) | 0.3 (2.58) | -2.9 (2.33) | 0.3 (1.95)
  Change from baseline in respiratory rate (breaths/minute) - Day 1, 1 hours post-dose | -0.8 (1.10) | -1.0 (1.58) | -1.8 (2.39) | -0.6 (1.71)
  Change from baseline in respiratory rate (breaths/minute) - Day 1, 4 hours post-dose | -0.8 (1.10) | 0.3 (1.77) | -1.1 (1.79) | 1.4 (2.32)
  Change from baseline in respiratory rate (breaths/minute) - Day 2 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in respiratory rate (breaths/minute) - Day 2 post-dose | -2.4 (1.67) |  |  |
  Change from baseline in respiratory rate (breaths/minute) - Day 3 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 3 post-dose |  | 0 (0) | -1.8 (3.08) | -1.1 (1.60)
  Change from baseline in respiratory rate (breaths/minute) - Day 4 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 4 post-dose |  | 0.1 (1.79) | 0 (0) | 0 (0)
  Change from baseline in respiratory rate (breaths/minute) - Day 7 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 7 post-dose |  | 0.1 (1.27) | -1.3 (1.73) | 0.1 (1.73)
  Change from baseline in respiratory rate (breaths/minute) - Day 8 post-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in respiratory rate (breaths/minute) - Day 8 post-dose | -2.4 (1.67) |  |  |
  Change from baseline in respiratory rate (breaths/minute) - Day 10 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 10 post-dose |  | 15.3 (1.41) | 0 (0) | 0 (0)
  Change from baseline in respiratory rate (breaths/minute) - Day 11 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 11 post-dose |  | 0 (0) | -1.6 (2.13) | 1.3 (2.16)
  Change from baseline in respiratory rate (breaths/minute) - Day 14 post-dose | -1.6 (0.89) | -1.1 (1.37) | -2.0 (2.45) | -1.3 (1.83)
  Change from baseline in respiratory rate (breaths/minute) - Day 28 post-dose: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in respiratory rate (breaths/minute) - Day 28 post-dose |  | -0.3 (2.00) | -1.6 (2.40) | -0.1 (1.85)

8. Primary Outcome: Changes From Baseline of Hematocrit.
Description: Clinical laboratory safety data will be summarized by laboratory measures such as hematocrit. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hematocrit (g/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Hematocrit (g/L)
  Change from baseline in hematocrit (L/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in hematocrit (L/L) Day 2 | 0.016 (0.0336) |  |  |
  Change from baseline in hematocrit (L/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hematocrit (L/L) Day 3 |  | 0 (0) | -0.010 (0.0211) | -0.008 (0.0217)
  Change from baseline in hematocrit (L/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hematocrit (L/L) Day 4 |  | -0.011 (0.0292) | 0 (0) | 0 (0)
  Change from baseline in hematocrit (L/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hematocrit (L/L) Day 7 |  | -0.006 (0.0167) | -0.031 (0.0169) | -0.016 (0.0232)
  Change from baseline in hematocrit (L/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in hematocrit (L/L) Day 8 | 0.006 (0.0270) |  |  |
  Change from baseline in hematocrit (L/L) Day 14 | 0.000 (0.0381) | -0.019 (0.0228) | -0.017 (0.0141) | -0.011 (0.0202)
  Change from baseline in hematocrit (L/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in hematocrit (L/L) Day 28 |  | -0.013 (0.0216) | -0.016 (0.0265) | 0.000 (0.0245)

9. Primary Outcome: Change From Baseline in Platelets (10^9/L)
Description: Clinical laboratory safety data will be summarized by laboratory measures such as platelets. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Platelets (10^9 cells/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Platelets (10^9 cells/L)
  Change from baseline in platelets (10^9/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in platelets (10^9/L) Day 2 | 2.0 (18.07) |  |  |
  Change from baseline in platelets (10^9/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in platelets (10^9/L) Day 3 |  | 0 (0) | -5.4 (18.87) | -7.3 (7.84)
  Change from baseline in platelets (10^9/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in platelets (10^9/L) Day 4 |  | -4.4 (12.67) | 0 (0) | 0 (0)
  Change from baseline in platelets (10^9/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in platelets (10^9/L) Day 7 |  | 0.9 (22.77) | -12.6 (10.86) | -9.2 (11.52)
  Change from baseline in platelets (10^9/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in platelets (10^9/L) Day 8 | 8.4 (16.64) |  |  |
  Change from baseline in platelets (10^9/L) Day 14 | -2.4 (27.65) | 15.9 (30.55) | 12.3 (25.74) | 21.2 (24.68)
  Change from baseline in platelets (10^9/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in platelets (10^9/L) Day 28 |  | 1.8 (34.30) | -11.2 (12.56) | 12.0 (39.31)

10. Primary Outcome: Change From Baseline in Neutrophils.
Description: Clinical laboratory safety data will be summarized by laboratory measures like neutrophils. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Neutrophils (10^9 cells/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Neutrophils (10^9 cells/L)
  Change from baseline in neutrophils (10^9/L) Day 2 | 0.56 (0.847) | 0 (0) | -0.33 (0.602) | 0.43 (0.817)
  Change from baseline in neutrophils (10^9/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in neutrophils (10^9/L) Day 3 |  | 0 (0) | -0.33 (0.602) | 0.43 (0.817)
  Change from baseline in neutrophils (10^9/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in neutrophils (10^9/L) Day 4 |  | 0.2 (0.555) | 0 (0) | 0 (0)
  Change from baseline in neutrophils (10^9/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in neutrophils (10^9/L) Day 7 |  | 0.36 (0.664) | -0.34 (1.181) | 2.06 (1.465)
  Change from baseline in neutrophils (10^9/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in neutrophils (10^9/L) Day 8 | -0.18 (0.536) |  |  |
  Change from baseline in neutrophils (10^9/L) Day 14 | -0.38 (0.838) | 0.27 (1.190) | -0.56 (0.932) | 0.13 (0.538)
  Change from baseline in neutrophils (10^9/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in neutrophils (10^9/L) Day 28 |  | 0.12 (0.653) | -0.62 (1.174) | 0.24 (0.855)

11. Primary Outcome: Change From Baseline of Alkaline Phosphatase.
Description: Clinical laboratory safety data will be summarized by laboratory measures such as alkaline phosphatase. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Alkaline Phosphatase (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Alkaline Phosphatase (U/L)
  Change from baseline in alkaline phosphatase (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in alkaline phosphatase (U/L) Day 2 | 2.2 (7.36) |  |  |
  Change from baseline in alkaline phosphatase (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alkaline phosphatase (U/L) Day 3 |  | 0 (0) | -0.9 (2.13) | -0.8 (2.39)
  Change from baseline in alkaline phosphatase (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alkaline phosphatase (U/L) Day 4 |  | -2.6 (3.06) | 0 (0) | 0 (0)
  Change from baseline in alkaline phosphatase (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alkaline phosphatase (U/L) Day 7 |  | 0.8 (8.18) | 2.1 (5.88) | -2.8 (4.61)
  Change from baseline in alkaline phosphatase (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in alkaline phosphatase (U/L) Day 8 | 1.8 (7.29) |  |  |
  Change from baseline in Alkaline Phosphatase (U/L) Day 14 | -1.8 (7.29) | -0.7 (9.29) | 1.2 (7.68) | -2.9 (4.43)
  Change from baseline in alkaline phosphatase (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alkaline phosphatase (U/L) Day 28 |  | -0.8 (3.79) | 7.0 (11.37) | 3.7 (8.9)

12. Primary Outcome: Change From Baseline in Alanine Transaminase.
Description: Clinical laboratory safety data will be summarized by laboratory measures like alanine transaminase. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Alanine Transaminase (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Alanine Transaminase (U/L)
  Change from baseline in alanine transaminase (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in alanine transaminase (U/L) Day 2 | -0.4 (2.30) |  |  |
  Change from baseline in alanine transaminase (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alanine transaminase (U/L) Day 3 |  | 0 (0) | -0.9 (2.13) | -0.8 (2.39)
  Change from baseline in alanine transaminase (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alanine transaminase (U/L) Day 4 |  | -2.6 (3.06) | 0 (0) | 0 (0)
  Change from baseline in alanine transaminase (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alanine transaminase (U/L) Day 7 |  | 0.8 (8.18) | 2.1 (5.88) | -2.8 (4.61)
  Change from baseline in alanine transaminase (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in alanine transaminase (U/L) Day 8 | -2.0 (2.24) |  |  |
  Change from baseline in alanine transaminase (U/L) Day 14 | 0.2 (2.24) | -0.7 (9.29) | 1.2 (7.68) | -2.9 (4.43)
  Change from baseline in alanine transaminase (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in alanine transaminase (U/L) Day 28 |  | -0.8 (3.79) | 3.7 (11.37) | 3.7 (8.90)

13. Primary Outcome: Change From Baseline in Asparate Aminotransferase.
Description: Clinical laboratory safety data will be summarized by laboratory measures like asparate aminotransferase. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Asparate aminotransferase (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Asparate aminotransferase (U/L)
  Change from baseline in asparate aminotransferase (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in asparate aminotransferase (U/L) Day 2 | -1.0 (5.24) |  |  |
  Change from baseline in asparate aminotransferase (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in asparate aminotransferase (U/L) Day 3 |  | 0 (0) | -0.8 (3.26) | -1.6 (2.5)
  Change from baseline in asparate aminotransferase (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in asparate aminotransferase (U/L) Day 4 |  | -2.1 (1.85) | 0 (0) | 0 (0)
  Change from baseline in asparate aminotransferase (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in asparate aminotransferase (U/L) Day 7 |  | 0.4 (5.50) | -2.2 (3.67) | -2.9 (5.99)
  Change from baseline in asparate aminotransferase (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in asparate aminotransferase (U/L) Day 8 | -1.0 (4.30) |  |  |
  Change from baseline in asparate aminotransferase (U/L) Day 14 | -0.4 (3.91) | 0.6 (6.95) | -3.7 (5.02) | -1.4 (4.40)
  Change from baseline in asparate aminotransferase (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in asparate aminotransferase (U/L) Day 28 |  | 1.2 (8.40) | 4.7 (16.73) | -0.1 (3.96)

14. Primary Outcome: Change From Baseline in Urea.
Description: Clinical laboratory safety data will be summarized by laboratory measures like urea. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Urea (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Urea (U/L)
  Change from baseline in urea (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in urea (U/L) Day 2 | -0.42 (0.740) |  |  |
  Change from baseline in urea (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in urea (U/L) Day 3 |  | 0 (0) | -0.25 (0.920) | -0.71 (1.746)
  Change from baseline in urea (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in urea (U/L) Day 4 |  | -0.27 (1.036) | 0 (0) | 0 (0)
  Change from baseline in urea (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in urea (U/L) Day 7 |  | 0.22 (1.018) | -0.54 (1.179) | -0.94 (0.840)
  Change from baseline in urea (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in urea (U/L) Day 8 | 0.24 (1.097) |  |  |
  Change from baseline in urea (U/L) Day 14 | -0.86 (1.167) | -0.28 (0.840) | -0.38 (1.232) | -0.56 (1.106)
  Change from baseline in urea (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in urea (U/L) Day 28 |  | 0.28 (1.272) | -0.20 (1.247) | -0.80 (1.103)

15. Primary Outcome: Change From Baseline in Creatinine.
Description: Clinical laboratory safety data will be summarized by laboratory measures like creatinine. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Creatinine (umol/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Creatinine (umol/L)
  Change from baseline in creatinine (umol/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in creatinine (umol/L) Day 2 | -2.8 (3.03) |  |  |
  Change from baseline in creatinine (umol/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in creatinine (umol/L) Day 3 |  | 0 (0) | 0.8 (4.73) | 1.0 (2.94)
  Change from baseline in creatinine (umol/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in creatinine (umol/L) Day 4 |  | -0.5 (7.01) | 0 (0) | 0 (0)
  Change from baseline in creatinine (umol/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in creatinine (umol/L) Day 7 |  | 0.7 (6.71) | -1.4 (6.42) | -1.7 (3.95)
  Change from baseline in Creatinine (umol/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in Creatinine (umol/L) Day 8 | 1.4 (3.78) |  |  |
  Change from baseline in creatinine (umol/L) Day 14 | -2.4 (7.54) | -1.3 (4.55) | -4.3 (5.81) | 1.6 (4.35)
  Change from baseline in creatinine (umol/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in creatinine (umol/L) Day 28 |  | 3.5 (7.37) | -4.4 (6.46) | -1.7 (6.63)

16. Primary Outcome: Change From Baseline in Gamma Glutamyl Transferase.
Description: Clinical laboratory safety data will be summarized by laboratory measures like gamma glutamyl transferase. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Gamma Glutamyl Transferase (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Gamma Glutamyl Transferase (U/L)
  Change from baseline in gamma glutamyl transferase (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in gamma glutamyl transferase (U/L) Day 2 | -0.6 (3.78) |  |  |
  Change from baseline in gamma glutamyl transferase (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in gamma glutamyl transferase (U/L) Day 3 |  | 0 (0) | -1.1 (1.97) | -0.1 (2.08)
  Change from baseline in gamma glutamyl transferase (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in gamma glutamyl transferase (U/L) Day 4 |  | -0.6 (2.91) | 0 (0) | 0 (0)
  Change from baseline in gamma glutamyl transferase (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in gamma glutamyl transferase (U/L) Day 7 |  | -0.7 (2.78) | -0.1 (2.32) | 1.0 (2.45)
  Change from baseline in gamma glutamyl transferase (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in gamma glutamyl transferase (U/L) Day 8 | -1.0 (2.55) |  |  |
  Change from baseline in gamma glutamyl transferase (U/L) Day 14 | 0.2 (1.48) | -0.3 (3.47) | 1.0 (3.67) | 0.4 (2.59)
  Change from baseline in gamma glutamyl transferase (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in gamma glutamyl transferase (U/L) Day 28 |  | -1.0 (2.62) | 2.2 (3.80) | 0.6 (3.10)

17. Primary Outcome: Change From Baseline in Bilirubin.
Description: Clinical laboratory safety data will be summarized by laboratory measures like bilirubin. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Bilirubin (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Bilirubin (U/L)
  Change from baseline in bilirubin (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in bilirubin (U/L) Day 2 | -1.0 (3.16) |  |  |
  Change from baseline in bilirubin (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in bilirubin (U/L) Day 3 |  | 0 (0) | 1.9 (2.92) | -0.5 (2.42)
  Change from baseline in bilirubin (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in bilirubin (U/L) Day 4 |  | 1.2 (1.87) | 0 (0) | 0 (0)
  Change from baseline in bilirubin (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in bilirubin (U/L) Day 7 |  | 0.6 (4.07) | -1.2 (4.15) | 2.1 (2.88)
  Change from baseline in bilirubin (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in bilirubin (U/L) Day 8 | -0.4 (3.51) |  |  |
  Change from baseline in bilirubin (U/L) Day 14 | -3.4 (3.21) | -0.1 (3.60) | -3.1 (2.32) | -0.1 (3.70)
  Change from baseline in bilirubin (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in bilirubin (U/L) Day 28 |  | 1.9 (3.60) | -1.9 (2.80) | -0.7 (3.83)

18. Primary Outcome: Change From Baseline in Lactate Dehydrogenase.
Description: Clinical laboratory safety data will be summarized by laboratory measures like lactate dehydrogenase. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Lactate Dehydrogenase (U/L)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Lactate Dehydrogenase (U/L)
  Change from baseline in Lactate Dehydrogenase (U/L) Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in Lactate Dehydrogenase (U/L) Day 2 | -0.8 (58.13) |  |  |
  Change from baseline in Lactate Dehydrogenase (U/L) Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in Lactate Dehydrogenase (U/L) Day 3 |  | 0 (0) | -7.4 (15.04) | -13.2 (14.80)
  Change from baseline in Lactate Dehydrogenase (U/L) Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in Lactate Dehydrogenase (U/L) Day 4 |  | -12.3 (26.24) | 0 (0) | 0 (0)
  Change from baseline in Lactate Dehydrogenase (U/L) Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in Lactate Dehydrogenase (U/L) Day 7 |  | -11.7 (32.39) | -25.7 (20.32) | -9.8 (21.44)
  from baseline in Lactate Dehydrogenase (U/L) Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  from baseline in Lactate Dehydrogenase (U/L) Day 8 | -14.4 (53.58) |  |  |
  Change from baseline in Lactate Dehydrogenase (U/L) Day 14 | -11.4 (65.22) | -7.5 (43.48) | -27.6 (22.39) | -3.7 (23.76)
  Change from baseline in Lactate Dehydrogenase (U/L) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in Lactate Dehydrogenase (U/L) Day 28 |  | -12.9 (41.15) | -16.4 (23.01) | -12.0 (19.20)

19. Primary Outcome: Change From Baseline of Prothrombin Intl. Normalized Ratio.
Description: Clinical laboratory safety data will be summarized by laboratory measures like prothrombin intl. normalized ratio. Observed values and changes from baseline for continuous clinical laboratory parameters will be summarized at each scheduled timepoint using descriptive statistics. Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. The clinical assessment of laboratory data will be summarized at each scheduled timepoint using participant counts and percentages. Individual participant profiles will be presented for any laboratory parameters with at least one post-dose value outside the laboratory's reference ranges that is deemed clinically significant.
Time Frame: For Part A on Days 2, 8 and 14 and For Part B on Days 3 or 4, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Prothrombin Intl. Normalized Ratio
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Prothrombin Intl. Normalized Ratio
  Change from baseline in prothrombin intl. normalized ratio Day 2: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in prothrombin intl. normalized ratio Day 2 | -0.06 (0.055) |  |  |
  Change from baseline in prothrombin intl. normalized ratio Day 3: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in prothrombin intl. normalized ratio Day 3 |  | 0 (0) | 0.01 (0.057) | -0.03 (0.048)
  Change from baseline in prothrombin intl. normalized ratio Day 4: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in prothrombin intl. normalized ratio Day 4 |  | 0.01 (0.032) | 0 (0) | 0 (0)
  Change from baseline in prothrombin intl. normalized ratio day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in prothrombin intl. normalized ratio day 7 |  | 0.02 (0.067) | 0.01 (0.033) | 0.00 (0.047)
  Change from baseline in prothrombin intl. normalized ratio Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in prothrombin intl. normalized ratio Day 8 | -0.02 (0.045) |  |  |
  Change from baseline in prothrombin intl. normalized ratio day 14 | -0.06 (0.055) | -0.01 (0.057) | 0.00 (0.050) | -0.02 (0.042)
  Change from baseline in prothrombin intl. normalized ratio Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in prothrombin intl. normalized ratio Day 28 |  | 0.00 (0.047) | 0.02 (0.044) | 0 (0)

20. Primary Outcome: Changes From Baseline of Single RR Heart Rate (Beats/Min).
Description: The following ECG parameters will be analyzed: single RR heart rate (beats/min). Observed values and changes from baseline for single RR heart rate (beats/min). will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: Change from baseline to Day 14 for the Sentinel Cohort (Part A), and change from baseline to Day 28 for the Main Cohort (Part B).
Population: The Sentinel Cohort (Part A) had their end of study visit at Day 14, while the Main Cohort (Part B) had their end of study visit at Day 28.
Measure: Mean (Standard Deviation); unit: Single RR heart rate (beats/min)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Single RR heart rate (beats/min)
  Change from baseline in single RR heart rate (beats/min) Day 14: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in single RR heart rate (beats/min) Day 14 | 5.00 (3.940) |  |  |
  Change from baseline in single RR heart rate (beats/min) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in single RR heart rate (beats/min) Day 28 |  | 3.08 (8.160) | 0.54 (6.610) | 2.29 (7.010)

21. Primary Outcome: Changes From Baseline of QRS Duration, Single Beat (ms).
Description: The following ECG parameters will be analyzed: QRS duration, single beat (ms). Observed values and changes from baseline for ECG parameters will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: QRS duration, single beat (ms)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
QRS duration, single beat (ms)
  Change from baseline in QRS duration (ms) Day 14: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in QRS duration (ms) Day 14 | 2.06 (4.210) |  |  |
  Change from baseline in QRS duration (ms) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in QRS duration (ms) Day 28 |  | 2.24 (2.780) | 0.38 (5.770) | -1.95 (5.170)

22. Primary Outcome: Change From Baseline in PR Interval, Single Beat (ms).
Description: The following ECG parameters will be analyzed: PR interval (ms). Observed values and changes from baseline for ECG parameters will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: PR Interval, single beat (ms)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
PR Interval, single beat (ms)
  Change from baseline in PR Interval, single beat (ms) Day 14: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in PR Interval, single beat (ms) Day 14 | -4.94 (12.880) |  |  |
  Change from baseline in PR Interval, single beat (ms) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in PR Interval, single beat (ms) Day 28 |  | -0.51 (6.870) | 1.06 (3.960) | -1.53 (11.380)

23. Primary Outcome: Change From Baseline in QTcB Interval, Single-beat (ms)
Description: The following ECG parameters will be analyzed: QTcB Interval. Observed values and changes from baseline for ECG parameters will be summarized at each scheduled timepoint using descriptive statistics.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: QTcB Interval, Single-beat (ms)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
QTcB Interval, Single-beat (ms)
  Change from baseline in QTcB Interval, Single-beat (ms) Day 14: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in QTcB Interval, Single-beat (ms) Day 14 | 0.78 (21.290) |  |  |
  Change from baseline in QTcB Interval, Single-beat (ms) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in QTcB Interval, Single-beat (ms) Day 28 |  | 4.08 (13.040) | -2.38 (13.380) | -1.44 (15.580)

24. Primary Outcome: Change From Baseline in QTcF Interval (ms).
Description: The following ECG parameters will be analyzed: QTcF Interval (ms). Observed values and changes from baseline for ECG parameters will be summarized at each scheduled timepoint using descriptive statistics.
  For QTcF Interval, the number of participants with values greater than 450 (and 480, 500) msec or an increase from baseline of at least 30 (and 60) msec will also be tabulated, in accordance with International Conference of Harmonization (ICH) E14
Time Frame: Change from baseline to end of study.
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: QTcF Interval (ms)
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
QTcF Interval (ms)
  Change from baseline in QTcF Interval (ms) Day 14: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in QTcF Interval (ms) Day 14 | -4.54 (17.810) |  |  |
  Change from baseline in QTcF Interval (ms) Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in QTcF Interval (ms) Day 28 |  | 0.92 (8.730) | -2.91 (14.320) | -3.47 (11.680)

25. Primary Outcome: Changes From Baseline Nasal Symptoms Using the Sino-Nasal Outcome Test (Total Score)
Description: The sino-nasal outcome test (SNOT-22) is to measure the consequences of rhinosinusitis. Scores will be totaled for all 22 items. The minimum score on the sinonasal outcome test-22 (SNOT-22) is 0 and the maximum score is 110. Changes from baseline in individual total sinonasal outcome test-22 (SNOT-22) scores will be calculated as the post-baseline value minus the baseline value. Thus, a negative change will reflect an improvement in the corresponding score. Observed values and changes from baseline will be summarized at each scheduled timepoint by treatment using descriptive statistics and tabulated for each cohort (dose level) and overall.
  Individual symptoms will be listed, with the 5 most important issues flagged. The total SNOT score will also be included in the listing.
Time Frame: For Part A Days 1 and 8. For Part B Days 1, 7, 14 and 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Sinonasal outcome test-22 scores
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
Number analyzed (Participants) | 5 | 10 | 9 | 10
Sinonasal outcome test-22 scores
  Change from baseline in SNOT-22 scores - Day 1 | 2.6 (4.83) | 1.9 (1.79) | 1.4 (2.17) | 1.1 (1.20)
  Change from baseline in SNOT-22 scores - Day 7: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in SNOT-22 scores - Day 7 |  | -1.0 (3.12) | -2.1 (4.29) | 3.4 (6.80)
  Change from baseline in SNOT-22 scores - Day 8: number analyzed (Participants) | 5 | 0 | 0 | 0
  Change from baseline in SNOT-22 scores - Day 8 | 2.4 (3.36) |  |  |
  Change from baseline in SNOT-22 scores - Day 14: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in SNOT-22 scores - Day 14 |  | 3.0 (10.54) | -3.0 (3.82) | 3.3 (7.47)
  Change from baseline in SNOT-22 scores - Day 28: number analyzed (Participants) | 0 | 10 | 9 | 10
  Change from baseline in SNOT-22 scores - Day 28 |  | 0.7 (7.82) | -3.6 (3.93) | -0.5 (2.32)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Sentinel Cohort | Main Cohort Group 1 | Main Cohort Group 2 | Main Cohort Group 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/5 | 9/10 | 10/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Cohort (N=5) | Main Cohort Group 1 (N=10) | Main Cohort Group 2 (N=10) | Main Cohort Group 3 (N=10)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 6 (7) | 3 (3) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 5 (5) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Viral upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4) | 3 (3)
Ansomnia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hyposmia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (8) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Nasuea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neotrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT06030414/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT06030414/SAP_001.pdf